CLINICAL TRIAL: NCT04839224
Title: Comparing Between CO2 and Phenylephrine Treatment in Patients With Progressive Lacunar Infarction (CARBOGEN Study)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow Patient Enrollment
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2020-1491
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Acute Ischemic Stroke
Keywords: CO2; carbogen; phenylephrine; lacunar infarction; progressive stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke, Lacunar | interventions — carbogen; Phenylephrine

STUDY DESIGN:
Intervention Model Description: 1. The study is a single center, prospective, randomized, open-label trial with blinded end-point assessment (PROBE) design study.
  2. For the patients with neurological worsening after lacunar infarction, the carbogen group and the phenylephrine group will be randomized by 1: 1.
  3. Patients will be enrolled from April 2021 to December 2022 (based on the date of stroke).
  4. We will collect medical history, laboratory findings, neurological scores, and functional recovery.
  5. Functional recovery scores are performed by independent researchers in the blind state.
  6. All data is collected using e-CRF, and the image study will be anonymized and sent to the central adjudication.
  7. Central adjudication will review the image study.
Who Masked: Outcomes Assessor
Masking Description: Three months after discharge, the independence assessment will be performed by the researcher who don't know the patients group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbogen group (Experimental)
  Interventions: Drug: carbogen
- Phenylephrine group (Active Comparator)
  Interventions: Drug: phenylephrine

INTERVENTIONS:
Drug: carbogen — Patients will inhale carbogen gas for 10 minutes and rest for 50 minutes.
  Arms: Carbogen group
Drug: phenylephrine — Start phenylephrine with 0.5 mg/hr and titrate upto 3.5 mg/hr or systolic blod pressure 200 mmHg.
  Arms: Phenylephrine group

SUMMARY:
Lacunar infarction is an ischemic stroke occurred by small perforating artery occlusion . Twenty percent of ischemic stroke is lacunar infarction.

However, outcome of lacunar infarction is excellent, about 20-40% patients are suffered neurological worsening.

Progressive lacunar infarction is associated poor functional outcome and neurological deficit.

Currently, no treatment for progressive lacunar infarction is recommended on the guideline.

Several small study reported that phenylephrine and magnesium may be helpful for progressive lacunar infarction.

Carbogen is a mixture of 5% CO2 with 95% O2. Carbogen is safe and it is used for the treatment of sudden sensory neural hearing loss or ocular ischemia.

CO2 dilate cerebral arteriole and concentration of CO2 is correlated with cerebral blood flow.

Lacunar infarction is small and perfused with marginal flow by neighboring perforating arteriole.

Increased cerebral blood flow following dilation of cerebral arteriole by CO2 might halt and revert progressive lacunar infarction.

Induced hypertension is alternative treatment of progressive lacunar infarction. Increasing blood pressure also induce cerebral blood flow.

Phenylephrine is an α1 agonist, phenylephrine act on peripheral artery and little effect on cerebral artery or heart.

Several studies reported that the effectiveness of phenylephrine on progressing stroke.

Therefore, this study will compare the effectiveness of carbogen versus phenylephrine in lacunar infarction patients who suffered neurological worsening.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥20 years
2. Anterior circulation progressive lacunar infarction.
3. Neurological worsening either 1 point in NIHSS score or MRC grade

Exclusion Criteria:

1. Age <20
2. Cortical infarction
3. Posterior circulation lacunar infarction
4. Relevant artery stenosis more than 50% or occlusion
5. Moyamoya disease
6. Difficulty in inhalation of Carbogen (panic, severe anxiety disorder)
7. Drug allergy for phenylephrine
8. Persistent bradycardia (pulse rate < 50 /min)
9. History of hemorrhagic stroke
10. Pre-stroke mRS ≥2

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
percent improvement of NIHSS score in each group | 48 hours
  (baseline NIHSS score-post-treatment NIHSS score)/baseline NIHSS score×100
difference of NIHSS score in each group | 48 hours
  baseline NIHSS score-post-treatment NIHSS score
percent improvement of MRC score in each group | within 48 hours
  (baseline MRC score-post-treatment MRC score)/baseline MRC score×100
difference of MRC score in each group | within 48 hours
  baseline MRC score-post-treatment MRC score
Safety outcome: Side effect | within 7 days
  Side effect (cerebral hemorrhage, myocardial infarction, Losing consciousness, difficulty breathing, dizziness, fatigue, headache, anxiety, etc)
Safety outcome: discontinuing patients | within 7 days
  Number of discontinuing patients due to side effects

SECONDARY OUTCOMES:
Comparison between groups by percent improvement of NIHSS score | 48 hours
  (baseline NIHSS score-post-treatment NIHSS score)/baseline NIHSS score×100
Comparison between groups by difference of NIHSS score | 48 hours
  baseline NIHSS score-post-treatment NIHSS score
Comparison between groups by percent improvement in MRC score | within 48 hours
  (baseline MRC score-post-treatment MRC score)/baseline MRC score×100
Comparison between groups by difference of MRC score | within 48 hours
  baseline MRC score-post-treatment MRC score
Functional independence | upon discharge, 3 months after onset
  modified Rankin score 0 to 2

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Suk Nam, MD, PhD, Principal Investigator — Department of Neurology, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No